CLINICAL TRIAL: NCT03168074
Title: A Phase II Window-of-opportunity Study of Single Agent Lenvatinib in Estrogen Receptor Positive Early Stage Breast Cancer
Brief Title: Phase II Study of Single Agent Lenvatinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Eisai Co., Ltd. (Industry); Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR02/07/16
Record Dates: First submitted 2017-03-26; First posted 2017-05-30 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Intervention Model Description: A Phase II window-of-opportunity study of single agent lenvatinib in estrogen receptor positive early stage breast cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lenvatinib (Experimental): Eligible patients will be treated with approximately 2 weeks of single agent lenvatinib (range 10-28 days, depending on the date of breast cancer surgery; last dose of lenvatinib to be administered no later than 48 hours before surgery in patients who are planned to receive ≤14 days lenvatinib, and no later than 120 hours before surgery in patients who are planned to receive 15-28 days lenvatinib).
  Interventions: Drug: lenvatinib

INTERVENTIONS:
Drug: lenvatinib — Eligible patients will be treated with approximately 2 weeks of single agent lenvatinib (range 10-28 days, depending on the date of breast cancer surgery; last dose of lenvatinib to be administered no later than 48 hours before surgery in patients who are planned to receive ≤14 days lenvatinib, and no later than 120 hours before surgery in patients who are planned to receive 15-28 days lenvatinib).Tissue sections from the pre-treatment and post-treatment tumor will be collected for biomarker analysis. Pre- and post-treatment ultrasound will be used to document the size of the target lesions.

SUMMARY:
The Investigators hypothesize that single agent lenvatinib has biological activity in estrogen receptor positive breast cancer, and that the effects are more pronounced in patients with positive RET expression in the tumor.

DETAILED DESCRIPTION:
Background and Rationale of Study:

A. RET and Endocrine Resistance in Breast Cancer RET is an estrogen response gene, and preclinical studies have demonstrated cross talk between RET and ER. Significant interactions between RET and ERα pathways have been described, with increased response to estrogen stimulation observed in the presence of functional RET. RET is associated with resistance to tamoxifen and aromatase inhibitors, and increased RET expression has been demonstrated in hormone resistant cell lines and primary tumors.Combined anti-estrogen and anti-RET therapy in luminal breast cancer had a greater effect on cell growth than either therapy alone. The two classes of drugs have different mechanisms of action; a RET TKI reduced growth through induction of apoptosis, while anti-ERα reduced cell proliferation, forming the biologic basis for dual treatment.Dual therapy with tamoxifen and vandetinib, a RET inhibitor, resulted in greater reduction in tumor growth rate in MCF7 xenografts in mice.RET has been reported to be over-expressed in up to 75% of ER+ breast cancers (n=20), compared to only 10% of ER-negative breast cancers (n=10) in a small study. Recently, the investigators tested 94 archival breast cancer specimens from the National University Hospital, Singapore and found RET over-expression (2-3+) to be present in 59% of ER negative breast cancers (n=39) and 62% of ER positive breast cancers (n=55)

There is limited clinical experience in combining RET inhibitors with endocrine therapy in breast cancer, with only one reported study using vandetanib. In this study, 127 post-menopausal metastatic breast cancer patients with hormone receptor-positive, bone-predominant disease, were randomized to fulvestrant alone versus fulvestrant combined with vandetanib. No differences in clinical benefit rate, progression-free survival, or overall survival, were noted between the two treatment groups. Vandetanib, however, is a less potent inhibitor of RET than lenvatinib. Lenvatinib has been granted orphan drug designation for thyroid cancer by the United States Food and Drug Administration in 2013, but is not being actively developed in breast cancer.

The investigators tested 9 ER+ breast cancer cell lines for RET expression using Western blot, and identified 4 with high expression (BT474, MB361, HCC1419, UACC812), 2 with normal expression (MCF7, CAMA1), and 3 with low expression (T47D, ZR-75-1, BT483). To evaluate the effects of combining lenvatinib with endocrine therapy in ER+ breast cancer cell lines with different RET expression, the investigators performed experiments using 6 cell lines, including 2 with high RET expression (BT474, MB361), 2 with normal RET expression (MCF7, CAMA1), and 2 with low RET expression (T47D, ZR-75-1). IC50 to tamoxifen and lenvatinib alone was established for each cell line, followed by combination therapy at 3 different doses for each drug. Cell apoptosis and proliferation was measured using caspase 3/7 and MTT assays respectively. Preliminary experiments showed lenvatinib to have activity in ER positive breast cancer cell lines, regardless of levels of RET expression. Lenvatinib was at least additive with tamoxifen in all 6 ER positive breast cancer cell lines tested, with the combination resulting in ≥50% cell kill compared to single agent tamoxifen in BT474, CAMA1, and T47D cell lines. These pre-clinical observations suggest the potential role of lenvatinib in combination with endocrine therapy in the treatment of ER positive breast cancers.

Cells were seeded on 96-well plates and after 24 hours, the cells were treated with tamoxifen and lenvatinib simultaneously at different doses (tamoxifen at 0, 1, or 5µM, lenvatinib at 0, 5, 10 µM) and incubated for 72 hours. Cell viability was assessed using CCK-8 assay.

B. Preliminary observation of clinical activity of single agent lenvatinib in hormone receptor positive breast cancer

The investigators previously hypothesized that combining a RET inhibitor such as lenvatinib with endocrine therapy may potentiate anti-tumor effects in hormone receptor positive breast cancers. The investigators have recently initiated a study of lenvatinib + letrozole as neoadjuvant therapy in hormone receptor positive breast cancer patients. Eligible patients were treated with two weeks of single agent lenvatinib, followed by 12 weeks of lenvatinib + letrozole. Two patients have been enrolled and the investigators observed tumor reduction of 10-15% on ultrasound after 2 weeks of single agent lenvatinib. To confirm these interesting observations, the investigators intend to treat a larger cohort of patients with newly diagnosed early stage breast cancer who are awaiting definitive breast cancer surgery with approximately 2 weeks of single agent lenvatinib using a window-of-opportunity design, and evaluate tumor response on ultrasound and histological changes from pre- and post-treatment tumor biopsies. This design will allow the investigators to expand the target population for rapid enrollment to achieve a quick signal on biological activity of lenvatinib in human breast cancers in vivo.

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfill ALL the following inclusion criteria

* Female ≥18 years
* Histological or cytological diagnosis of breast carcinoma
* No prior treatment for current breast carcinoma
* Scheduled for upfront definitive breast cancer surgery (breast conserving surgery or mastectomy with or without sentinel lymph node biopsy or axillary lymph node clearance)
* Estrogen receptor positive (>1%)
* Adequate bone marrow, renal and liver function
* Adequate organ function including the following:

  * Bone marrow:

    * Absolute neutrophil (segmented and bands) count (ANC) >= 1.5 x 109/L
    * Platelets >= 100 x 109/L
  * Hepatic:

    * Bilirubin < = 1.5 x upper limit of normal (ULN),
    * ALT or AST < = 2.5x ULN, (or < = 5 X with liver metastases)
  * Renal:

    * Creatinine < = 1.5x ULN
* Normal thyroid function
* Able to swallow pills
* Able to sign informed consent
* Able to comply with study-related procedures

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons:

* Scheduled for neoadjuvant systemic therapy
* Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Treatment within the last 28 days with any investigational drug.
* Major surgery within 28 days of study drug administration.
* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Poorly controlled diabetes mellitus.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment
* Symptomatic brain metastasis.
* History of significant neurological or mental disorder, including seizures or dementia.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is designed for breast cancer patients. Male breast cancer is extremely rare and we do not intend to include this rare population.
Enrollment: 30 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2021-03-28 (Estimated); Study Completion 2021-03-28 (Estimated)

PRIMARY OUTCOMES:
Biological effects of short-course single agent lenvatinib in estrogen receptor positive breast cancer using a window-of-opportunity design | after 10-28 days of single agent lenvatinib
  To evaluate Ki67 changes. The Ki-67 protein is a cellular marker for proliferation. It is strictly associated with cell proliferation. Ki67 has been shown to be a surrogate marker of biological activity and treatment response in estrogen receptor positive breast cancer treated with endocrine therapy.
Biological effects of short-course single agent lenvatinib in estrogen receptor positive breast cancer using a window-of-opportunity design | after 10-28 days of single agent lenvatinib
  To evaluate histological response such as the improvement in the appearance of microscopic tissue specimens after treatment with lenvatinib. The improved appearance of biopsy specimens after treatment often suggests the patient's prognosis will improve as well.
Biological effects of short-course single agent lenvatinib in estrogen receptor positive breast cancer using a window-of-opportunity design | after 10-28 days of single agent lenvatinib
  To evaluate apoptosis. Apoptosis is the death of cells which occurs as a normal and controlled part of an organism's growth or development. The presence of apoptosis indicates anti-cancer effects.
Biological effects of short-course single agent lenvatinib in estrogen receptor positive breast cancer using a window-of-opportunity design | after 10-28 days of single agent lenvatinib
  To evaluate RET. RET is an estrogen response gene. RET is associated with resistance to tamoxifen and aromatase inhibitors, and increased RET expression has been demonstrated in hormone resistant cell lines and primary tumors.
Biological effects of short-course single agent lenvatinib in estrogen receptor positive breast cancer using a window-of-opportunity design | after 10-28 days of single agent lenvatinib
  To evaluate downstream targets such as AKT. AKT /protein kinase B (PKB) is a cardinal node in diverse signaling cascades important in both normal cellular physiology and various disease states. AKT signaling regulates cell proliferation and survival, cell growth (size), glucose metabolism, cell motility and angiogenesis. Aberrant regulation of these processes results in cellular perturbations considered hallmarks of cancer, and numerous studies testify to the frequent hyperactivation of AKT signaling in many human cancer.
Biological effects of short-course single agent lenvatinib in estrogen receptor positive breast cancer using a window-of-opportunity design | after 10-28 days of single agent lenvatinib
  To evaluate downstream targets such as ERK. ERK is Extracellular signal-regulated kinase. Deregulation of ERK signalling pathway is linked to many other aspects of the tumour phenotype.

SECONDARY OUTCOMES:
Changes in the primary tumor dimensions | after 10-28 days of single agent lenvatinib
  to obtain the percentage change in primary breast tumor dimension measured by ultrasound
The proportion of subjects with tumor reduction | after 10-28 days of single agent lenvatinib
  to obtain the proportion of subjects with tumor reduction of at least 10%
Comparison of the clinical response of lenvatinib in RET negative versus RET positive, ER positive breast cancers | after 10-28 days of single agent lenvatinib
  To compare clinical response of lenvatinib in RET negative versus RET positive, ER positive breast cancers
Comparison in the overall average changes in biological effects of lenvatinib between RET negative and RET positive, ER positive breast cancers. | after 10-28 days of single agent lenvatinib
  : Comparison of the number of patients with Ki67 changes, histological response, apoptosis, RET and downstream targets such as AKT and ERK, between RET negative versus RET positive, ER positive breast cancers.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, Principal Investigator — National University Hospital, Singapore; Ching Wan Chan, Principal Investigator — National University of Singapore; Ern Yu Tan, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Nationa University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boulay A, Breuleux M, Stephan C, Fux C, Brisken C, Fiche M, Wartmann M, Stumm M, Lane HA, Hynes NE. The Ret receptor tyrosine kinase pathway functionally interacts with the ERalpha pathway in breast cancer. Cancer Res. 2008 May 15;68(10):3743-51. doi: 10.1158/0008-5472.CAN-07-5100. PMID 18483257
- [Background] Plaza-Menacho I, Morandi A, Robertson D, Pancholi S, Drury S, Dowsett M, Martin LA, Isacke CM. Targeting the receptor tyrosine kinase RET sensitizes breast cancer cells to tamoxifen treatment and reveals a role for RET in endocrine resistance. Oncogene. 2010 Aug 19;29(33):4648-57. doi: 10.1038/onc.2010.209. Epub 2010 Jun 7. PMID 20531297
- [Background] Morandi A, Martin LA, Gao Q, Pancholi S, Mackay A, Robertson D, Zvelebil M, Dowsett M, Plaza-Menacho I, Isacke CM. GDNF-RET signaling in ER-positive breast cancers is a key determinant of response and resistance to aromatase inhibitors. Cancer Res. 2013 Jun 15;73(12):3783-95. doi: 10.1158/0008-5472.CAN-12-4265. Epub 2013 May 6. PMID 23650283